CLINICAL TRIAL: NCT04365036
Title: A Multicenter, Phase 3, Randomized Trial of Sequencial Chemoradiotherapy with or Without Toripalimab (PD-1 Antibody) in Newly Diagnosed Early-Stage Extranodal Natural Killer/T Cell Lymphoma, Nasal Type (ENKTL)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qingqing Cai, Chief physician, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2020-040-01
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: NK/T Cell Lymphoma Nos
MeSH Terms: interventions — toripalimab; pegaspargase; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- toripalimab with P-GemOx (Experimental): Patients will receive toripalimab and induction chemotherapy with pegaspargase, gemcitabine, oxaliplatin, every 3 weeks for 4 cycles before radiation. Definitive intensity-modulated radiotherapy (IMRT) will be given. Concurrent toripalimab of 240mg will be administered every 3 weeks for 3 cycles during IMRT. Toripalimab 240mg will be given every 3 weeks for 13 cycles, started on day 1 of induction chemotherapy.
  Interventions: Drug: Toripalimab; Drug: Pegaspargase; Drug: Gemcitabine; Drug: Oxaliplatin; Radiation: Definitive intensity-modulated radiotherapy (IMRT)
- P-GemOx (Active Comparator): Patients will receive induction chemotherapy with pegaspargase, gemcitabine, oxaliplatin, every 3 weeks for 4 cycles before radiation. Definitive intensity-modulated radiotherapy (IMRT) will be given.
  Interventions: Drug: Pegaspargase; Drug: Gemcitabine; Drug: Oxaliplatin; Radiation: Definitive intensity-modulated radiotherapy (IMRT)

INTERVENTIONS:
Drug: Toripalimab — toripalimab 240mg, d1, intravenous drip
  Arms: toripalimab with P-GemOx
Drug: Pegaspargase — pegaspargase, 2000U/m2, d1, intravenous drip
Drug: Gemcitabine — gemcitabine, 1000mg/m2, d1,d8, intravenous drip
Drug: Oxaliplatin — oxaliplatin, 130mg/m2, d1, intravenous drip,
Radiation: Definitive intensity-modulated radiotherapy (IMRT) — Definitive intensity-modulated radiotherapy (IMRT) of 54-56Gy will be given in 25~26 days

SUMMARY:
The purpose of this randomized, multi-center,phase Ⅲ clinical trail is to compare the safety and efficacy of sequencial chemoradiotherapy with or without toripalimab (PD-1 antibody) for newly diagnosed early-stage extranodal natural killer/T-cell lymphoma, nasal type (ENKTL)

ELIGIBILITY:
Inclusion Criteria:

* biopsy proved extranodal natural killer/T-cell lymphoma, nasal type;
* newly diagnosed stage I/II patients;
* at least one evaluable lesion；
* ECOG PS 0-2;
* 18-75 years; without other malignancy;
* proper functioning of the major organs.

Exclusion Criteria:

* hemophagocytic syndrome or aggressive NK cell leukemia;
* involvement of central nervous system;
* previously received treatment of chemotherapy, radiotherapy, immunotherapy or biotherapy for lymphoma；

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Estimated)
Dates: Start 2020-05-03 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
progression free survival (PFS) | 3 years

SECONDARY OUTCOMES:
complete remission (CR) rate | From the start of treatment with the interventions until 6 months
overall response rate (ORR) | From the start of treatment with the interventions until 6 months
overall survival (OS) | 3 years
recurrence-free survival (RFS) | 3 years
event free survival (EFS) | 3 years
disease-free survival (DFS) | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong General Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No